CLINICAL TRIAL: NCT04370964
Title: Evolution of Family Alliance in Families With a Designated Adolescent Patient (12-18 Years) During a Family Therapy Process: Prospective Pilot Study
Brief Title: Evolution of Family Alliance in Families With a Designated Adolescent Patient (12-18 Years) During a Family Therapy Process
Acronym: LTP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, Januel, Psychiatrist, head of the clinical research department, Centre hospitalier de Ville-Evrard, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10477M-LTP
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Family Relations
Keywords: family alliance-family relionship-co-parenting-Lausanne Trilogy Play LTP

STUDY DESIGN:
Intervention Model Description: The family will be evaluated in two stages via the standardized situations LTP (parents and patient) and LFP (family) as well as self-assessments, before the start of the therapy then after 9 months of therapy, each family being its own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family with young aged people (Other): The family will be evaluated in two stages via the standardized situations LTP (parents and patient) and LFP (family) as well as self-assessments
  Interventions: Other: Lausanne Trilogy Play; Other: Lausanne Family Play

INTERVENTIONS:
Other: Lausanne Trilogy Play — Trilogical game of Lausanne ("Lausanne Trilogue Play" in English abbreviated LTP), which allows an evaluation of the family alliance. This systematic observation provides a "snapshot" of the family structure and its adaptive abilities. It is based on the assumption that the ability to solve "small" tasks is representative of the ability to solve more important tasks.The LTP consists of modelling the different possibilities of interaction in a triad according to a four-part scenario: 1) one parent plays with the child, the other parent is simply present; 2) the parents switch roles; 3) both parents play together with the child; and 4) both parents have to talk together.
  Other Names: LTP
Other: Lausanne Family Play — Lausanne Family Play (LFP) is a game situation adapted to families with more than one child. Thus, like the LTP, the LFP takes place in four phases:1) one parent plays with siblings while the other is in a third-observer position; 2) the parents reverse their roles;3) children play while parents are talking and 4) family members play together.
  Other Names: LFP

SUMMARY:
The proposed study focuses on the relational characteristics of the family and their evolution in the course of family therapy, through the evolution of the family alliance (degree of coordination achieved by its members to perform a task) and co-parenting (support that the mother and father give each other in their roles as parents), assuming that the family therapy allows the improvement of these two aspects. The family alliance is evaluated via a standardized observation situation (Lausanne Family Play LFP adapted from the Lausanne Trilogy Play LTP) whose sessions are filmed. The alliance assessment is carried out by the coding and scales of the FASS (Family Alliance Assessment Scales,) tool during viewing.

ELIGIBILITY:
Inclusion Criteria:

* Families attended in family therapy by the G02 sector teams and the Bondy family therapy team attached to G14 and I05, with a designated adolescent patient (aged 12-18).
* Family whose parents or co-parents live under the same roof. Co-parents designate adults to be responsible for the care and education of one or more children (Talbot &Mchale, 2004)
* Blended families

Exclusion Criteria:

* Single parent family without co-parents (in-laws, grandparents...) living under the same roof
* Insufficient mastery of French
* Separated parents (lack of daily life is unsuitable for scales chosen)
* patient without social security scheme
* Persons in emergency situations.
* Persons unable to give their personal consent, of whom adults under guardianship

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2021-03-05 (Estimated); Study Completion 2021-09-05 (Estimated)

PRIMARY OUTCOMES:
Family Alliance Assessment Sales (FASS) | Between "month 1" and "month 3"
  Scale validated in French evaluating the family alliance when viewing Lausanne Trilogy Play
Family Adaptability and Cohesion Evaluation Scales for adolescents(FACES III) | At baseline
  It consists of 40 items: a questionnaire for adolescents (40 items) . It was designed to make it possible to "make a relational diagnosis" on the family and to bridge the gap between theory, research and practice in family psychology, based on the three dimensions that make up the "circomplexe" model.
Family Adaptability and Cohesion Evaluation Scales for adolescents (FACES III) | at month "9"
  It consists of 40 items: a questionnaire for adolescents (40 items) . It was designed to make it possible to "make a relational diagnosis" on the family and to bridge the gap between theory, research and practice in family psychology, based on the three dimensions that make up the "circomplexe" model.
Family Adaptability and Cohesion Evaluation Scales for parents (FACES III) | At Baseline
  It consists of 40 items: a questionnaire for parents (40 items). It was designed to make it possible to "make a relational diagnosis" on the family and to bridge the gap between theory, research and practice in family psychology, based on the three dimensions that make up the "circomplexe" model.
Family Adaptability and Cohesion Evaluation Scales for parents (FACES III) | at month "9"
  It consists of 40 items: a questionnaire for parents (40 items). It was designed to make it possible to "make a relational diagnosis" on the family and to bridge the gap between theory, research and practice in family psychology, based on the three dimensions that make up the "circomplexe" model.
The Coparenting Inventory for Parents and Adolescents (CI-PA) | At Baseline
  Validated in English, this scale was translated into French by the Favez team and is used by the Lausanne team for their LTP protocol with adolescents. This is a Self Questionnaire of 38 items for the teenager and 25 items for the parents.
The Coparenting Inventory for Parents and Adolescents (CI-PA) | At month "9"
  Validated in English, this scale was translated into French by the Favez team and is used by the Lausanne team for their LTP protocol with adolescents. This is a Self Questionnaire of 38 items for the teenager and 25 items for the parents.
Family Attitude Scale, l'échelle d'attitude familiale (FAS-30) | At baseline
  This questionnaire concerns thoughts and emotions that family members may have towards each other and is intended to assess the degree of hostility of the parent towards the patient. Each item is rated according to its frequency, ranging from 4 (daily) to 0 (never). There are 20 "negative" items (they refer to the parent's criticism of the patient and the burden they feel because of the patient) and 10 "positive" items (the patient's affection and positive feelings).
Family Attitude Scale, l'échelle d'attitude familiale (FAS-30) | At month 9
  This questionnaire concerns thoughts and emotions that family members may have towards each other and is intended to assess the degree of hostility of the parent towards the patient. Each item is rated according to its frequency, ranging from 4 (daily) to 0 (never). There are 20 "negative" items (they refer to the parent's criticism of the patient and the burden they feel because of the patient) and 10 "positive" items (the patient's affection and positive feelings).
Child Behavior Check List (CBCL) | at baseline
  The CBCL is the most widely used questionnaire by researchers in the field of children's development and behaviour. The CBCL has been translated and validated in several languages and intercultural studies have shown its relevance and richness. It is validated and translated into French. There is an adaptation for the school age group 6-18 years.
Child Behavior Check List (CBCL) | at month 9
  The CBCL is the most widely used questionnaire by researchers in the field of children's development and behaviour. The CBCL has been translated and validated in several languages and intercultural studies have shown its relevance and richness. It is validated and translated into French. There is an adaptation for the school age group 6-18 years.

SECONDARY OUTCOMES:
Security in the inter parental subsystem: le questionnaire de sécurité dans le sous- système parental (SIS). | At baseline
  Validated in English and reproduced and translated into French by Francesco Lopez and Favez Nicolas, this is a self-assessment for the teenager (43 Items) to evaluate the "emotional security system".
Security in the inter parental subsystem: le questionnaire de sécurité dans le sous- système parental (SIS). | At month 9
  Validated in English and reproduced and translated into French by Francesco Lopez and Favez Nicolas, this is a self-assessment for the teenager (43 Items) to evaluate the "emotional security system".

OTHER OUTCOMES:
Mchale Co-parenting Scale | at baseline
  The French version of this parent self-assessment is validated and includes 16 questions plus a preliminary question (Frascarolo F, 2009) Depending on the questions they are asked, parents are sometimes asked to think about when they are with their spouse and child and sometimes when they are alone with their child. They must estimate the frequency of certain behaviours.
Mchale Co-parenting Scale | at month 9
  The French version of this parent self-assessment is validated and includes 16 questions plus a preliminary question (Frascarolo F, 2009) Depending on the questions they are asked, parents are sometimes asked to think about when they are with their spouse and child and sometimes when they are alone with their child. They must estimate the frequency of certain behaviours.
Dyadic Adjustment Scale (DAS) | at baseline
  This is a scale widely used in research, validated in French (Antoine et al, 2008).
  It is composed of 16 items that explore two dimensions of the conjugal relationship: -the first dimension concerns the "degree of agreement in the couple", it is composed of 10 items relating to areas of divergence (divorce, annoyance) or convergence (common goals, joint attitude in relations with the environment). There are also items of affective expression, consensus and satisfaction. -The second dimension consists of six items and corresponds to the "quality of the dyadic interactions": the domains and the behaviors of exchange and partnership in the couple.
Dyadic Adjustment Scale (DAS) | at month 9
  This is a scale widely used in research, validated in French (Antoine et al, 2008).
  It is composed of 16 items that explore two dimensions of the conjugal relationship: -the first dimension concerns the "degree of agreement in the couple", it is composed of 10 items relating to areas of divergence (divorce, annoyance) or convergence (common goals, joint attitude in relations with the environment). There are also items of affective expression, consensus and satisfaction. -The second dimension consists of six items and corresponds to the "quality of the dyadic interactions": the domains and the behaviors of exchange and partnership in the couple.
The questionnaire on the developmental stages of families | at baseline
  This is a questionnaire developed by Marie France Bradley and Robert Pauzé.It was conceived according to the developmental hypothesis of the family, which must, throughout its life cycle, go through a number of stages, namely: the departure from the house of the young single adult, the formation of the couple, the arrival of the children, the entry of children into adolescence, the departure of children from the family, the retirement of parents. For each of these steps, the family needs to reorganize. This instrument seeks to assess whether the developmental tasks they face have been carried out with more or less difficulty.
The questionnaire on the developmental stages of families | at month 9
  We decided to pass only the part about the family with teenagers. This part contains 43 items, corresponding to developmental tasks divided into 7 categories (support for the autonomy and responsibility of the adolescent, redefining the power of the parents vis-à-vis the adolescent, support for socialisation, support for the identity and personal development of the adolescent, impact of adolescence on the parental couple, multiple demands in adolescence and new issues in adolescence).

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Christine Beaucousin, MBBS, Principal Investigator — CHVille Evrard
Locations (1):
- EPS Ville Evrard, Aubervilliers, France

IPD SHARING:
Plan to Share IPD: Undecided